CLINICAL TRIAL: NCT00913276
Title: Conditioning With Volatile Anesthetics in Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University Ghent (Other); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: StV 15-2008
Record Dates: First submitted 2009-05-27; First posted 2009-06-04 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: End-stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane anesthesia (Other)
  Interventions: Drug: Sevoflurane
- Propofol anesthesia (Other)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol
  Arms: Propofol anesthesia
Drug: Sevoflurane
  Arms: Sevoflurane anesthesia

SUMMARY:
The gap between the number of candidates for orthotopic liver transplantation and the availability of suitable liver grafts has led to a rise in deaths on most waiting lists. Strategies applied in many centers to minimize this deficit include living donation or split of a cadaveric organ for two recipients, domino transplantation, and the use of so-called expanded criteria donors. Alternatively, conditioning of an organ would also allow protec-tion of the liver upon ischemia-reperfusion injury, possibly decreasing postoperative liver function and im-proving clinical outcome. The technique of conditioning with the volatile anesthetic sevoflurane is an easily applicable procedure which could be performed in any center worldwide.

Data and experience with sevoflurane attenuating ischemic-reperfusion injury in liver resection lead to the hypothesis of a beneficial effect of volatile anesthetics in liver transplantation. In this randomized controlled trial, patients will be randomly assigned to liver transplantation with propofol anesthesia (propofol group) or sevoflurane conditioning with the volatile anesthetic (sevoflurane group). Primary endpoint is postoperative peak of the transaminase (AST), secondary endpoints are complications, primary liver graft function, ICU and hospital stay. We hypothesis that patients with conditioning have an attenuated increase of transaminases as well as a better outcome.

ELIGIBILITY:
Inclusion criteria:

* Older than 18 years
* Patients undergoing liver transplantation
* Total or partial cadaveric liver transplantation
* Living related liver transplantation

Exclusion criteria:

* Patients unable to understand the German or Italian language
* Patients with known or suspected allergy to propofol, soja or egg
* Patients with norepinephrine infusion above 15 microg/min
* Intensive care patients with severe impairment of renal or pulmonary function (e.g. dialysis, hemofiltration, FiO2>0.5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-01; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
postoperative paek of AST | 4 y

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Beck Schimmer, Prof MD, Principal Investigator — University Hospital Zurich, Division of Anaesthesiology
Locations (1):
- University Hospital Zurich, Division of Anaesthesiology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Beck-Schimmer B, Bonvini JM, Schadde E, Dutkowski P, Oberkofler CE, Lesurtel M, DeOliveira ML, Figueira ER, Rocha Filho JA, Auler JO Jr, D'Albuquerque LA, Reyntjens K, Wouters P, Rogiers X, Debaerdemaeker L, Ganter MT, Weber A, Puhan MA, Clavien PA, Breitenstein S. Conditioning With Sevoflurane in Liver Transplantation: Results of a Multicenter Randomized Controlled Trial. Transplantation. 2015 Aug;99(8):1606-12. doi: 10.1097/TP.0000000000000644. PMID 25769076